CLINICAL TRIAL: NCT01113255
Title: Validation of a Simulated Clinical Evaluation of Ventilators
Acronym: SIMULVENTI
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P070146
Record Dates: First submitted 2010-02-26; First posted 2010-04-29 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-11

CONDITIONS: Respiratory Diseases; Chronic and Acute Respiratory Failure
Keywords: VENTILATORS; BENCH EVALUATION; MECHANICAL VENTILATION
MeSH Terms: conditions — Respiratory Tract Diseases; Bronchiolitis Obliterans Syndrome | interventions — Respiration, Artificial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHRONIC REPIRATORY FAILURE (Active Comparator)
  Interventions: Procedure: bench-evaluation, of three ventilators
- ACUTE RESPIRATORY FAILURE (Active Comparator)
  Interventions: Procedure: bench-evaluation, of three ventilators

INTERVENTIONS:
Procedure: bench-evaluation, of three ventilators — to select in-VITRO the most appropriate ventilator for a given pathology.
  Other Names: Mechanical ventilation

SUMMARY:
The purpose of this study is to evaluate the ability of a device reproducing patients' respiratory characteristics to select in-VITRO the most appropriate ventilator for a given pathology.

DETAILED DESCRIPTION:
Context : Mechanical ventilation is an essential element in the management of chronic as well as acute respiratory failure allowing an improvement of both mortality and morbidity. However, considering the wide choice of ventilators available on the market, it has become increasingly difficult to choose the most appropriate ventilator according to the pathology presented by a patient, patients being able to try only a limited number of devices. Patient-ventilator synchronization is a crucial part of ventilation efficacy and its success. It depends on both the physiopathological characteristics of patients and specific properties of the ventilation device.

Objective : To evaluate the ability of a device reproducing patients' respiratory characteristics to select in-VITRO the most appropriate ventilator for a given pathology.

Method : Multi-center transversal study. Selection, after an initial bench-evaluation, of three ventilators. Clinical evaluation of their efficacy and synchronization between patient and ventilator and establishment of a classification.

Second bench evaluation of the studied ventilators while the bench is simulating the ventilation characteristic of previously studied patients in order to compare the results obtained in VITRO to the results obtained in vivo.

Selection criteria : Patients requiring mechanical ventilation for management of either chronic or acute respiratory failure.

Patients, centers : 4 groups of 14 patients presenting chronic respiratory disease followed in the ICU of RAYMOND POINCARE HOSPITAL in GARCHES and in the pulmonary departments of the Armand Trousseau hospital and the PITIE SALPETRIERE IN PARIS; 1 cohort of 12 patients admitted in the ICU of Henri Mondor in CRETEIL IN PARIS for acute respiratory failure.

Study duration : 33 months (bench study : 3 + 6 months, clinical study : 24 months) Perspectives : Developing an evaluation tool allowing the rapid assessment of any new available ventilator according to the specific characteristics (and needs) of a patient and to a given pathology. Selecting the most appropriate ventilator for a given patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring mechanical ventilation for management of either chronic or acute respiratory failure.
* Old of at least 6 years
* Having given his consent writes after enlightened information, him even and the parents for least than 18 years, only he for most than 18 years
* Realization of a preliminary medical examination

Exclusion Criteria:

* Patients presenting criteria of pointed exacerbation of the respiratory disease

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2009-03; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Selection, after an initial bench-evaluation, of three ventilators. Clinical evaluation of their efficacy and synchronization between patient and ventilator and establishment of a classification. | 24 MONTHS

SECONDARY OUTCOMES:
Second bench evaluation of the studied ventilators while the bench is simulating the ventilation characteristic of previously studied patients in order to compare the results obtained in VITRO to the results obtained in vivo. | 24 MONTHS

CONTACTS AND LOCATIONS:
Overall Officials: Hélène Prigent, ph, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Raymond Poincaré, Garches, France